CLINICAL TRIAL: NCT07383350
Title: Improving Patient-centered Communication and Antibiotic Use With Information Sheets for Acute Respiratory Tract Infections: Study Protocol for a Pragmatic Cluster Randomized Trial in Danish General Practice (INFO-ARTI).
Brief Title: Improving Patient-centered Communication and Antibiotic Use With Information Sheets for Acute Respiratory Tract Infections: A Study Protocol
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Research Unit for General Practice in Aalborg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 471-2
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Acute Bronchitis; ACUTE SINUSITIS; Sore Throat
Keywords: Acute respiratory tract infections; Antibiotics; General practice; Patient-centered communication; Information sheets
MeSH Terms: conditions — Bronchitis; Pharyngitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care arm (No Intervention)
- ARTI Info-sheets (Active Comparator)
  Interventions: Other: ARTI Info-sheets

INTERVENTIONS:
Other: ARTI Info-sheets — ARTI Info-sheets are three information sheets design to be used together with patients contacting general practice with symptoms of acute respiratory tract infections. The information sheets is created as a dialog-tool to increase patient involvement in managing of acute respiratory tract infections.
  Arms: ARTI Info-sheets

SUMMARY:
The goal of this trial is to investigate if the use of information sheets regarding acute respiratory tract infections will lead to more rational antibiotic prescribing and increase patient-centered communication i Danish general practice.

The main questions to be answered:

* Will the use of information sheets lower antibiotic prescribing.
* Will the use of information sheets increase patient-centered communication.

We will compare use of information sheets in the consultation with patients with symptoms of acute respiratory tract infections to usual care (control) to find out if information sheets lower antibiotic prescribing.

Participants will be presented to the information sheets during the consultation regarding symptoms of acute respiratory tract infection.

Participants will fill in a short questionaire regarding patient-centered communication shortly after the consultation.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients must contact the general practice clinic with symptoms of either acute pharyngotonsillitis, acute rhinosinusitis or acute bronchitis and should be above 18 years of age.

Exclusion Criteria:

* Prior antibiotic treatment for the current episode of acute respiratory tract infections.
* Urgent need of hospitalization.
* Patients who do not understand Danish.
* Patients not listed within the general practice clinic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1144 (Estimated)
Dates: Start 2026-01-05 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients contacting the general practice clinic with symptoms of acute respiratory tract infections prescribed antibiotics at initial consultation. | At Initial consultation (day 0)

SECONDARY OUTCOMES:
Proportion of patients contacting the general practice clinic with symptoms of acute respiratory tract infections with redeemed antibiotic prescriptions within 14 days after the initial consultation. | Additional contact from day 0 until day 14.
Proportion of patients contacting the general practice clinic with symptoms of acute respiratory tract infections with retrieval of prescribed antibiotics from the pharmacy within 14 days after the initial consultation. | Retrieval of prescribed antibiotic from day 0 until day 14
Proportion of patients contacting the general practice clinic with symptoms of acute respiratory tract infections reconsultation within 14 days after the initial consultation. | Reconsultation from day 0 until day 14.
Proportion of patients contacting the general practice clinic with symptoms of acute respiratory tract infections with "out of hours"-consultations within 14 days after the initial consultation. | Out of hours consultation from day 0 until day 14.
Proportion of patients contacting the general practice clinic with symptoms of acute respiratory tract infections with hospital admissions within 14 after the initial consultation. | Hospital admissions from day 0 until day 14.
Proportion of patients experiencing high level of Patient-centered communication measured by CollaboRATE. | Day 0.

OTHER OUTCOMES:
Proportion of patients with one of the ARTI Info-sheets used during the consultation, as reported by healthcare professional. | At Initial consultation (day 0)
Proportion of patients where the ARTI info-sheets were meaningful to use, as reported by healthcare professional. | At Initial consultation (day 0)
Estimated additional meantime spent on consultation, when using ARTI Info-sheets, reported by healthcare professional. | At Initial consultation (day 0)

CONTACTS AND LOCATIONS:
Locations (1):
- Research Unit for General Practice in Aalborg, Aalborg, Denmark